CLINICAL TRIAL: NCT04565262
Title: Multi-center Study of IFN Combined With Nucleosides Analog Antiviral Therapy in Pediatric Patients With HBeAg Positive Chronic Hepatitis B (CHB) Aged 1-16 Years
Brief Title: Study on Antiviral Therapy for HBeAg-positive Chronic Hepatitis B Patients Aged 1-16 Years
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R2020050DA010
Record Dates: First submitted 2020-06-22; First posted 2020-09-25 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-08

CONDITIONS: HBeAg Positive Chronic Hepatitis B
Keywords: hepatitis B,chronic; Interferon ; Nucleosides;child
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Intervention Model Description: These subjects will be randomized (1:1) to group A(treated with NAs + IFN for 96 weeks) and group B(treated with NAs for 48 weeks, then NAs combined with IFN for 96 weeks).Meanwhile, 1-6 years and 7-16 years patients should be distributed by 1:1 ratio by random method in both groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAs+IFN-α (Experimental): NAs+IFN-α/ 96w
  Interventions: Drug: NAs+IFN-α
- NAs+(IFN-α+ NAs ) (Other): NAs/48w+(IFN-α+ NAs)/96w
  Interventions: Drug: NAs+IFN-α

INTERVENTIONS:
Drug: NAs+IFN-α — NAs+IFN-α:(NAs +IFN)/96 weeks：NAs（when the CHB patients<2years old, the drug is LAM）combined with IFN-α（when the CHB patients<3years old, the drug is IFN-α）for 96 weeks。 NAs+(NAs+IFN-α) :NAs/48weeks+(NAs+ IFN)/96 weeks：NAs（when the CHB patients<2years old, the drug is LAM）for 48 weeks ，then combined with IFN-α（when the CHB patients<3years old, the drug is IFN-α）for 96weeks。 Response guided treatment（RGT） by HBsAg quantification： The course of interferon alpha was 24 weeks after HBsAg and HBeAg turned negative up to 96 weeks, and NAs was discontinued 12 months after HBsAg serological conversion.

SUMMARY:
The purpose of this study is to provide theoretical and real world evidence for the optimization of antiviral treatment by IFN combined with Nucleosides analog in HBeAg positive chronic hepatitis B patients aged 1-16 years，so that the functional cure could be achieved in the greatest extent in pediatric patients

DETAILED DESCRIPTION:
This research is a national multicenter, randomized, prospective study. The planned sample size is 200 subjects in 1-16 years pediatric patients with HBeAg positive Chronic Hepatitis B (CHB). These subjects will be randomized (1:1) to group A(treated with NAs + IFN for 96 weeks) and group B(treated with NAs for 48 weeks, then NAs combined with IFN for 96 weeks).Meanwhile, 1-6 years and 7-16 years patients should be distributed by 1:1 ratio by random method in both groups. Regularly Blood cell count, biochemical test, hepatitis B viral markers test, and lymphocyte subsets test were exerted. To compare the curative effect of group A and group B, The primary monitoring indicator is HBsAg clearance rate, and the secondary monitoring indicator is hepatitis B virus (HBV) DNA clearance，HBeAg seroconversion in these patients,. So that we can make the optimal antiviral treatment strategy for 1-16-year-old children with CHB，and try to find out the possible influencing factors of function cure

ELIGIBILITY:
Inclusion Criteria:

1. Aged 1 to 16 years old.
2. Chronic Hepatitis B (CHB) patients or HBsAg positive > 6 months patients who are line with the diagnostic criteria for chronic hepatitis B infection.
3. ALT:40～400 U/L.
4. HBeAg positive.
5. HBV DNA>2×104IU/L.
6. Liver histology: G<3.
7. Agree to sign the Informed Consent Form (Children aged 1-6 years may be signed by the guardian; children between the ages of 7 and 11 are in principle signed by the child and the guardian; those over the age of 12 must be signed by the child and the guardian)

Exclusion Criteria:

1. white blood cell (WBC)< 3.5×109/L，PLT< 80×1012/L，Pt A<60%，total bilirubin (TBIL)>34umol/L，ALB<35g/L，Cr>133umol/L.
2. Combined with HAV、HCV、HDV、HEV or HIV-infected persons.
3. Patients combined with other causes of liver disease：alcoholic or non-alcoholic liver disease，thyroid disease，autoimmune liver disease，genetic metabolic liver disease，bile duct diseases，or Parasitic infection of hepatobiliary tract.
4. Patients with decompensated cirrhosis，including ascites.
5. Received the following medications（Immunosuppressant and Systemic cytotoxic drugs）in six months.
6. Patients who are allergy to IFNs and NAs;
7. Patients with other severe or active psychosomatic diseases （kidney, heart, lungs, vascular, neurological, digestive including history of pancreatitis, metabolic diseases including diabetes, thyroid and Adrenal disease, adrenal disease or tumor), Researchers believe which affect the treatment, evaluation or compliance of patients with the study plan.
8. Patients who unable to comply with the study arrangement judged by researcher.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
The rates of HBsAg serological disappearance / conversion in CHB patients at 48 weeks | 48 weeks
  The rates of HBsAg serological disappearance / conversion in CHB patients at 48 weeks
The rates of HBsAg serological disappearance / conversion in CHB patients at 96 weeks | 96 weeks
  The rates of HBsAg serological disappearance / conversion in CHB patients at 96 weeks
The rates of HBsAg serological disappearance / conversion in CHB patients at 144 weeks | 144 weeks
  The rates of HBsAg serological disappearance / conversion in CHB patients at 144 weeks
The rates of HBsAg serological disappearance / conversion in CHB patients at 168 weeks | 168 weeks
  The rates of HBsAg serological disappearance / conversion in CHB patients at 168 weeks

SECONDARY OUTCOMES:
The rate of HBeAg clearance / seroconversion | 168 weeks
  The rate of HBeAg clearance / seroconversion in patients with CHB
HBV DNA negative conversion rate | 168 weeks
  HBV DNA negative conversion rate in patients with CHB
ALT(Alanine aminotransferase) recovery rate | 168 weeks
  ALT recovery rate in patients with CHB

OTHER OUTCOMES:
Number of participants with treatment-related side effect and safety events as assessed by GSI | 168 weeks
  Side effect and safety events include adverse events, adverse drug reactions etc. during the treatment
Average duration of HBeAg seroconversion | 168 weeks
  Average duration of HBeAg seroconversion during treatment
Average duration of disappearance of HBsAg | 168 weeks
  Average duration of disappearance of HBsAg during treatment
Assessed the changes of liver stiffness measure by FibroScan after antiviral therapy | 168 weeks
  Comparison the changes of liver stiffness before and after antiviral treatment (evaluated by FibroScan)
Rate of relapse in patients after stop of antiviral therapy of NAs | 168 weeks
  Rate of relapse in patients after stop of antiviral therapy of NAs

CONTACTS AND LOCATIONS:
Overall Officials: Min Zhang, Dcotor, Principal Investigator — Beijing 302 Hospital
Locations (1):
- Min Zhang, Beijing, Beijing Municipality, China